CLINICAL TRIAL: NCT00479323
Title: Stimulation of Donors for Pneumococcal Reference Serum
Brief Title: Pneumococcal Reference Standard
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-0093
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2011-04

CONDITIONS: Pneumococcal Infections
Keywords: pneumococcal vaccine, Pneumovax, reference sera, serum 89SF
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

ARMS (1):
- 1 (Other): Immunize healthy volunteers with pneumococcal vaccine (Pneumovax 23) to obtain a pool of hyperimmune sera in a quantity sufficient to generate reference sera.
  Interventions: Biological: Pneumovax 23

INTERVENTIONS:
Biological: Pneumovax 23 — Licensed pneumococcal vaccine (Pneumovax 23).

SUMMARY:
Serum 89 SF is a supply of serum that was collected from people who were vaccinated with the pneumococcal vaccine in the late 1980s. The supply of this serum is running low. The purpose of this study is to give the pneumococcal vaccine to healthy volunteers and take serum blood samples in order to increase the reference serum supply. Study participants will include 250 healthy men and women, ages 18-45. Study procedures will include a physical exam, interviews, blood samples and blood testing. All volunteers will receive the pneumococcal vaccine in the deltoid muscle of the arm. Participants will be involved in the study for approximately 17 weeks.

DETAILED DESCRIPTION:
Serum 89SF is a pooled sera from individuals vaccinated with a 23 valent pneumococcal polysaccharide vaccine collected in the late 1980s. The 89SF standard for ELISA is running low (2-3 year supply) and is insufficient to serve for opsinophagocytosis assay (OPA), which requires large volumes. The objective of this study is to immunize healthy volunteers with licensed polyvalent pneumococcal polysaccharide vaccine (Pneumovax 23) with subsequent blood donation in a quantity sufficient to make reference sera. Two hundred fifty volunteer subjects will be recruited from a total population of up to 600. Study participants will include healthy men and nonpregnant females, ages 18-45. Subjects will undergo physical examination by a licensed clinician, subject interview, and clinical laboratory and serologic testing. Potential subjects must provide written informed consent and meet all eligibility criteria. On Day 0, subjects will receive 0.5 mL pneumococcal vaccine (Pneumovax 23) in the deltoid muscle. Volunteers will remain in the clinic for 30 minutes following immunization for observation of any adverse reactions. Volunteers will return to clinic in 10-35 days following immunization to donate 1 unit (approximately 500 mL) of blood. Volunteers will return for a second donation of 1 unit of blood not less than 8 weeks and not more than 14 weeks following the first donation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female between the ages of 18 to 45 and weighing a minimum of 110 pounds.
2. Women of childbearing potential (not surgically sterile or postmenopausal for >/= 1 year) must agree to practice adequate contraception (ie, barrier method, abstinence, intrauterine device, or licensed hormonal method) for the entire period while on protocol.
3. Women of childbearing potential must have a negative urine pregnancy test within 24 hours prior to vaccination and prior to each blood collection.
4. Participants must be afebrile and in general good health in the opinion of the investigator as determined by vital signs, medical history, and physical examination.
5. Subject laboratory tests, including hemoglobin, hematocrit, total white blood count and platelets, aspartate aminotransferase, alanine aminotransferase, and serum protein. All values must be within normal limits (WNL) except AST and ALT that must less than or equal to 1.5 X ULN and total serum protein >=6.0 gms; Males: hemoglobin >=13.5 gm/dL, hematocrit >=41% Females: hemoglobin >=12.5 gm/dL, hematocrit >=38%
6. Serology for hepatitis B (core antibody), C, HIV, rapid plasma reagin, immunoglobulin and HIV must be negative.
7. Subjects must have adequate venous access.
8. Participants must communicate an understanding of the protocol and provide written informed consent for the protocol.

Exclusion Criteria:

1. Has received any investigational drug or vaccine within the past 6 months or is currently in any phase of another clinical trial or intends to participate in another clinical trial in the next 6 months.
2. Has received any licensed inactivated vaccine within 2 weeks or licensed live vaccine within 4 weeks of screening.
3. Has a known allergy to any component of the Pneumovax 23 vaccine.
4. Has a history of receiving human blood or any derivative of human blood within the preceding 12 months.
5. Has no evidence of skin infection at the potential phlebotomy sites or evidence of systemic or generalized disease that could create a risk of contamination of the serum.
6. Has no history of viral hepatitis after the 11th birthday and no history of close contact with an individual diagnosed with viral hepatitis within the past year.
7. Is immunosuppressed as a result of underlying illness or treatment or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
8. Long-term use of oral or parenteral steroids or high-dose inhaled steroids within the past 6 months.
9. Has a diagnosis of schizophrenia, bipolar disease, major psychiatric diagnosis, or has ever been hospitalized for a psychiatric illness.
10. Has a history of alcohol or drug abuse in the past 5 years.
11. Has any acute or chronic condition that, in the opinion of the investigator, would render vaccination or blood donation unsafe or the participant unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To immunize healthy volunteers with pneumococcal vaccine (Pneumovax 23) to obtain a pool of hyperimmune sera in a quantity sufficient to generate reference sera. | Duration of study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States